CLINICAL TRIAL: NCT00421837
Title: Pilot Study of the Genotypic Analysis of Patients Infected With Influenza Virus Compared With Uninfected Spouse/Close Contact Controls
Brief Title: Pilot Study of Genotypic Analysis
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 06-0092; N01AI80007C
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2011-04

CONDITIONS: Influenza
Keywords: influenza, flu, genotypic analysis, sub-study
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sera and saliva

GROUPS / COHORTS (2):
- controls: household and other close contacts
- cases: elderly (>55) subjects hospitalized with Influenza

SUMMARY:
Influenza (the flu) is a leading cause of respiratory (breathing) illness that leads to sickness and death during the winter months. A better understanding of why certain people get the flu or get sicker with the flu than other people is important for developing improved vaccines and treatments. This study will look at the genetic makeup (determines each person's specific characteristics and traits) of 50 patients, older than 50, who were hospitalized with flu at Vanderbilt University during the 2006-2007 flu season. Their genetic makeup will be compared with the genetic makeup of 50 people who are not related but were in close daily contact with the flu patient and were not infected with flu virus. The study staff will collect a blood sample (contains genetic material) from each participant (flu patients and their contacts) for comparison. Flu patients will have completed a health survey as part of the previous study, and their contacts will complete a shorter version of this survey.

DETAILED DESCRIPTION:
Influenza is a leading vaccine preventable cause of respiratory illness that leads to substantial morbidity and mortality during the winter months. It is defined by a rapid-onset systemic illness, with patients presenting with fever, chills, cough, myalgias, headache and sore throat. Given the huge health burden caused by influenza and the ever present threat of a future pandemic, a better understanding of population genetic variation and its association with severe outcomes from influenza infection is critical for developing improved vaccines and treatments for the entire population of at risk persons. This study is a single-center, specimen collection pilot protocol designed to compare the genotype of patients, aged greater than 50 years, who are hospitalized with respiratory symptoms or fever at Vanderbilt University with culture or PCR confirmed influenza virus infection with individuals who are not related but are in close daily contact with the subject and are not infected with influenza virus during the 2006 - 2007 influenza season. This study is linked to DMID protocol 06-0051. All subjects will be recruited from those subjects who have been enrolled in Division of Microbiology and Infectious Diseases (DMID) parent study 06-0051, a Vaccine and Treatment Evaluation Units (VTEU)-funded respiratory disease surveillance study conducted during the 2006 - 2007 influenza season. If the subject has completed the surveillance parent study, (DMID study 06-0051), then he/she must have agreed to be contacted for future studies on the surveillance consent prior to enrollment into this sub-study. Controls for this study will be recruited via the index cases. This study will enroll 100 subjects total, 50 study subjects and 50 control subjects. The 50 study subjects will include individuals hospitalized with respiratory symptoms or fever and infected with influenza virus. The 50 control subjects will be uninfected, non-related individuals living in the same household or in close daily contact with the subject. The study staff will obtain 15 ml venous blood sample from each subject for genotyping studies. Subjects will have completed a health assessment as part of the parent trial and controls will be asked a shorter version of this survey which includes items such as: demographics, chronic disease history, history of immunosuppressive drugs or conditions, vaccination history, smoking history, and living conditions. The primary objectives of the study are to conduct whole genome array analysis on individuals with confirmed influenza virus infection and to compare their genotype with individuals who were likely exposed to influenza due to close daily contact, but are not genetically related.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged greater than or equal to 50 years
2. For SUBJECTS: Enrolled in a Vaccine Treatment and Evaluation Unit (VTEU)-funded surveillance study conducted during the 2006 - 2007 influenza season [Division of Microbiology and Infectious Diseases (DMID) study 06-0051]
3. Residents of surveillance areas
4. For SUBJECTS: Persons who have been hospitalized with respiratory symptoms or fever and polymerase chain reaction (PCR) or culture confirmed influenza virus OR
5. For CONTROLS: Living with or in frequent contact with SUBJECT
6. For CONTROLS: Genetically unrelated to the SUBJECT
7. Willing and able to provide signature documentation of informed consent or parental permission

Exclusion Criteria:

1. For SUBJECTS: Not enrolled in a Vanderbilt led respiratory disease surveillance study [Division of Microbiology and Infectious Diseases (DMID) study 06-0051]
2. For SUBJECTS: Receipt of blood products in the past 6 months
3. Anything in the opinion of the Investigator that would prevent the subject from successfully participating in this study
4. For CONTROLS: Influenza infection during the 2006-2007 flu season

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects > 55 yo hospitalized with Influenza vs healthy household members and close contacts
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
phenotypic analysis | at analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee, United States